CLINICAL TRIAL: NCT00232050
Title: Study of Omalizumab in Moderate to Severe Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025A1304
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Asthma
Keywords: Asthma, IgE, Omalizumab
MeSH Terms: conditions — Asthma; Epilepsy, Idiopathic Generalized | interventions — Omalizumab

INTERVENTIONS:
Drug: Omalizumab

SUMMARY:
This study will evaluate the safety and efficacy of omalizumab up to 16 weeks in adult patients with moderate to severe bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

* Allergic asthma patients
* Inadequately controlled patients

Exclusion Criteria:

* - History of severe anaphylactoid or anaphylactic reactions
* Previous treatment with omalizumab
* History of cancer or cancer

Other protocol-defined exclusion criteria may apply

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2002-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Morning peak expiratory flow (PEF) at baseline and end of treatment.

SECONDARY OUTCOMES:
Pulmonary function parameters measured by spirometer
Frequency of rescue medication use
Symptom score
Activities of daily living score
Nighttime sleep score

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Study Chair — Novartis Pharmaceuticals Japan